CLINICAL TRIAL: NCT03042585
Title: Phase I Study of Autologous Transplant Conditioned by Dose-Escalated Total Body Irradiation (TBI) and Standard Doses of Cyclophosphamide and Palifermin (Kepivance) for High Risk Non-Hodgkins Lymphoma
Brief Title: Autologous Transplant Using Dose-Escalated Total Body Irradiation & Cyclophosphamide & Palifermin for NHL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Patrick Stiff, MD and Director of Cardinal Bernardin Cancer Center, Loyola University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 108993
Record Dates: First submitted 2017-01-04; First posted 2017-02-03 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Relapsed Non Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma
Keywords: BMT; NHL; Non-Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma; Refractory Non-Hodgkin Lymphoma; autologous stem cell transplantation
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Whole-Body Irradiation

STUDY DESIGN:
Intervention Model Description: Dose-Escalated Total Body Irradiation (TBI) of 4 levels. Palifermin (Kepivance) is being supplied by the sponsor and is FDA approved to decrease the incidence and duration of severe oral mucositis in participants with hematologic malignancies who receive high doses of chemotherapy and radiation therapy followed by stem cell rescue.
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dose Level 1 (Experimental): The participants will receive Palifermin on Day -10, -9 and -8. Total Body Irradiation 1.64 Gy per Fraction for a total of 8 Fractions. The total amount would be 13.12 Gy. The participants will receive total body irradiation twice a day for four days (Day -7, -6, -5, and Day -4). Over the following two days, the participants will receive cyclophosphamide (Day -3 and -2). The participants will receive stem cell infusion on Day 0 and G-CSF given daily until engraftment occurs. Participants will receive Palifermin on Day 0, +1 and +2.
  Interventions: Radiation: Total body irradiation
- Dose Level 2 (Experimental): The participants will receive Palifermin on Day -10, -9 and -8. Total Body Irradiation 1.76 Gy per Fraction for a total of 8 Fractions. The total amount would be 14.08 Gy. The participants will receive total body irradiation twice a day for four days (Day -7, -6, -5, and Day -4). Over the following two days, the participants will receive cyclophosphamide (Day -3 and -2). The participants will receive stem cell infusion on Day 0 and G-CSF given daily until engraftment occurs. Participants will receive Palifermin on Day 0, +1 and +2.
  Interventions: Radiation: Total body irradiation
- Dose Level 3 (Experimental): The participants will receive Palifermin on Day -10, -9 and -8. Total Body Irradiation 1.88 Gy per Fraction for a total of 8 Fractions. The total amount would be 15.04 Gy. The participants will receive total body irradiation twice a day for four days (Day -7, -6, -5, and Day -4). Over the following two days, the participants will receive cyclophosphamide (Day -3 and -2). The participants will receive stem cell infusion on Day 0 and G-CSF given daily until engraftment occurs. Participants will receive Palifermin on Day 0, +1 and +2.
  Interventions: Radiation: Total body irradiation
- Dose Level 4 (Experimental): The participants will receive Palifermin on Day -10, -9 and -8. Total Body Irradiation 2.00 Gy per Fraction for a total of 8 Fractions. The total amount would be 16 Gy. The participants will receive total body irradiation twice a day for four days (Day -7, -6, -5, and Day -4). Over the following two days, the participants will receive cyclophosphamide (Day -3 and -2). The participants will receive stem cell infusion on Day 0 and G-CSF given daily until engraftment occurs. Participants will receive Palifermin on Day 0, +1 and +2.
  Interventions: Radiation: Total body irradiation

INTERVENTIONS:
Radiation: Total body irradiation — When radiation is given in a way to cover the whole body, it is called total body irradiation.

SUMMARY:
Most participants with a relapsed or refractory non-Hodgkin's lymphoma that receive an autologous transplant are likely to suffer a relapse because standard myeloablative preparative regimens are unable to produce a cure. The majority of these participants do not have a stem cell donor available, are too frail to undergo an allogeneic transplant, or refuse an allograft. Historically these participants with high risk non-Hodgkin's lymphoma have had a very poor outcome.

To take advantage of the low transplant related mortality associated with an autologous transplantation, the investigators propose modifying the preparative regimen to make it more effective without increasing toxicity. By increasing the dose of radiation while administering the protective growth factor palifermin (Kepivance), the investigators hope to decrease the risk of relapse without increasing transplant related mortality.

Three prospective randomized trials have studied different radiation schemes as a part of the TBI and cytoxan preparative regimen prior to allogeneic transplantation for patients with AML or CML. As a group these trials showed that higher doses of TBI in these older studies decreased the risk of relapse at the expense of VOD, GVHD, and CMV. Three retrospective studies have also postulated that higher dose radiation led to less risk of relapse.

DETAILED DESCRIPTION:
This is a non-randomized, open-label phase I trial in participants with non-Hodgkin's lymphoma. The preparative regimen will be as follows:

Day -10 (prior to transplant) Palifermin treatment to prevent mouth sores Day -9 Palifermin treatment to prevent mouth sores Day -8 Palifermin treatment to prevent mouth sores Day -7 Total Body Irradiation twice a day Day -6 Total Body Irradiation twice a day Day -5 Total Body Irradiation twice a day Day -4 Total Body Irradiation twice a day Day -3 Cytoxan chemotherapy infusion Day -2 Cytoxan chemotherapy infusion Day -1 Day of rest Day 0 Stem cell infusion (bone marrow transplant), Palifermin treatment to prevent mouth sores and G-CSF given daily until stem cells take hold (engraftment) occurs.

Day +1 Palifermin treatment to prevent mouth sores Day +2 Palifermin treatment to prevent mouth sores

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* Participants scheduled to undergo autologous stem cell transplantation with relapsed or refractory non-Hodgkin's Lymphoma with less than a partial remission to salvage therapy.
* Participants scheduled to undergo autologous stem cell transplantation with relapsed or refractory non-Hodgkin's Lymphoma with any site of disease 2 cm or greater on pre-transplant imaging.
* Participants must have a performance status (PS) of 0-1.
* Participants must have acceptable kidney function.
* Acceptable pulmonary function test of the lungs.
* Acceptable liver function tests.

Exclusion Criteria:

* Participants must not have cutaneous T-cell, mantle cell, or lymphoblastic lymphoma.
* Participants must not have prior peripheral blood or marrow transplantation.
* Participants must not have prior radiation.
* Participants must not have significant history of uncontrolled cardiac disease; for example, uncontrolled hypertension, unstable angina, recent myocardial infarction (within prior 6 months), uncontrolled congestive heart failure, and cardiomyopathy with decreased ejection fraction.
* Participants must not have active bacterial, fungal, or viral infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Determine the frequency and severity of adverse events by evaluating grade 3 and grade 4 adverse events. | 4 weeks
  Any grade 3 or 4 dose limiting toxicities as described : • Heart failure with only minor response to medical therapy
  * Hemorrhagic cystitis with frank blood requiring sclerosing agent or other surgical procedure
  * Acute kidney failure requiring dialysis
  * Interstitial pneumonitis requiring ventilatory support or FiO2 > 50% x 24hrs
  * Bilirubin > 20 mg/dL
  * Unexplained seizures or coma
  * Severe mucositis requiring intubation for airway protection
  * Ileus requiring nasogastric decompression.
  * Death

SECONDARY OUTCOMES:
Blood work will be used to evaluate recovery of white blood cells, red blood cells and platelets. | 4 weeks
  To evaluate labwork during treatment and for 28 days post treatment
Pulmonary Function Test will be used to evaluate side effects of total body irradiation | 1 year
  Pulmonary Function Test will be used to evaluate side effects of total body irradiation.
CT scan or physical exam will be used to evaluate progression free survival. | 1 year
  CT scan or physical exam will be used to evaluate progression free survival as deemed necessary.
Mucositis measured by investigators. | At the start of treatment and daily until mucositis resolves or 28 days post transplant whichever comes first.
  Mucositis physical examination done by investigators by accessing the mouth using the WHO (World Health Organization) oral toxicity scale.
Number of participants with Grade 4 through 5 Adverse Events that are related to study treatment, grading according to NCI CTCAE Version 3. | 28 days post treatment
  Dose-limiting toxicities that are probably or definitely related to the treatment regimen.
Mucositis measured by oral mucositis questionnaires | At the start of treatment and daily until mucositis resolves or 28 days post transplant whichever comes first.
  The participants will complete the oral mucositis daily questionnaires prior to the physical assessment. The questionnaire includes the participants self-reported mouth and throat soreness.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Stiff, MD, Principal Investigator — Loyola University
Locations (1):
- Patrick Stiff, MD, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No